CLINICAL TRIAL: NCT01071356
Title: Intensive Motivational Interviewing for Methamphetamine Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Public Health Institute, California (Other)
Responsible Party: Principal Investigator, Alcoholresearchgroup, Douglas L Polcin, Ed.D, Public Health Institute, California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01DA024714 (NIH)
Record Dates: First submitted 2010-02-17; First posted 2010-02-19 (Estimated); Results first posted 2018-05-24 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-04

CONDITIONS: Methamphetamine Dependence
Keywords: methamphetamine; motivational interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive MI (Experimental): 9 hours of Motivational Interviewing + outpatient substance abuse treatment
  Interventions: Behavioral: Intensive MI
- Single session MI (Active Comparator): 1.5 hours of Motivational Interviewing + 8 hours of time equivalent nutrition classes +outpatient substance abuse treatment
  Interventions: Behavioral: Single session MI

INTERVENTIONS:
Behavioral: Intensive MI — Weekly individual therapy sessions over 9 weeks (Intensive MI condition) consisting of supportive and directive interventions. The control condition consists on a single session of MI and nutritional education.
  Arms: Intensive MI
Behavioral: Single session MI — Comparator arm that includes 1.5 hours of MI, 8 hours of nutrition classes and outpatient substance abuse treatment
  Arms: Single session MI

SUMMARY:
A Stage 2 randomized clinical trial (RCT) to test the efficacy of a 9-session model of motivational interviewing (MI) for methamphetamine (MA) dependence. Stage 1 pilot testing indicated the intervention could be easily learned and implemented with fidelity. The tailored treatment approach draws upon our previous conceptual papers on MI as well as our experience with a variety of MI protocols, including two Clinical Trials Network (CTN) studies of MI. An innovative feature of the "Higher Dose Motivational Enhancement Therapy" manual is that it comprehensively addresses the issues of clients who have achieved sustained sobriety as well as those still using substances. Thus, it is designed to facilitate treatment entry and engagement as well as maintenance of the gains made in treatment. MA dependent clients (N=220) were recruited from New Leaf outpatient treatment in Lafayette, California. Study participants were randomly assigned to 1) a single session of Motivational Interviewing (MI) plus 8 hours of health/nutrition education, or 2) the intensive 9-session MI intervention. In addition to the study interventions, both groups received standard outpatient treatment services at New Leaf. Study participants were assessed weekly during the first 9 weeks of treatment for MA use. More extensive assessments were conducted at treatment entry and 2-, 4-and 6-month follow-ups. Two therapists were "crossed" to treat clients in both conditions. Primary outcome measures included Timeline Follow Back (TLFB) for MA use, MA urinalysis results, and retention in treatment. Secondary outcomes include Addiction Severity Index scales and the TLFB for alcohol and other drugs. A mediation model will build upon MI research proposed by Moyers (2005) and our construct of "supportive confrontation" by testing whether feedback enhanced with warnings about the potential harm of MA use facilitates the therapeutic alliance, and whether this in turn facilitates better outcome. Clients with MA dependence are good candidates for a more intensive dose of MI because of their severe medical and psychosocial problems.

DETAILED DESCRIPTION:
This proposal responds to PA-07-111, "Behavioral & Integrative Treatment Development Program" issued by the National Institute on Drug Abuse. Based on promising pilot data, we propose to test the efficacy of a 9-session Motivational Interviewing (MI) manual for treating methamphetamine (MA) dependence (Galloway, Polcin, Kielstein, Brown & Mendelson, 2007; Polcin, Galloway, Palmer & Mains, 2004; Polcin, Brown & Galloway, 2005). (See Appendix A for a copy of the Intensive and Standard Manuals and Appendix B for our papers describing the rationale for its structure). The study builds upon a progression in our work from initial conceptualization of a more intensive model of MI (Polcin, et al., 2004), to development of the "Higher Dose Motivational Enhancement Therapy Manual" (Polcin, et al., 2005), to presentation of very promising stage 1 pilot data (Galloway, et al, 2007). The proposed study represents a logical next step in this research program.

In a meta-analysis of MI studies, Burke, Arkowitz & Menchola (2003) found that higher doses of MI were associated with better outcome. Based on this finding, they called for new studies to compare the effectiveness of standard low dose and more intensive MI. This proposal responds to that call. To date, no direct comparisons between high and low intensity MI have been published, and we are not aware of any intensive manuals other than the one presented here.

Our proposal addresses the aims of the NIDA Program Announcement (PA-07-111) well because the announcement calls for innovations and refinements of behavioral therapies for understudied populations. Clients with MA dependence are specifically identified as an understudied population in need of behavioral therapy trials. MA use is rampant in the Western U.S. and is growing in other parts of the country as well as oversees (Anglin et al., 2007; Rawson & Condon, 2007). Studies have shown MA dependent individuals frequently present serious medical and psychiatric conditions that complicate treatment efforts (Rawson, et al., 2000, 2004). Based on excellent retention of clients during our pilot testing (see Pilot Study outcomes in the Preliminary Studies section), we hypothesize intensive MI will be particularly useful in improving high treatment dropout rates and low engagement among MA dependent clients. Behavioral interventions are particularly needed because there are currently no evidence based pharmacological protocols for treating MA dependence (Vocci & Appel, 2007).

In this proposal, our "standard" MI condition is a single session of manual based MI (Martino et al., 2006) plus eight hours of health/nutrition education using a structured educational format (Harris, 2003, 2006). A copy of both MI interventions can be found in Appendix A and a draft version of the nutrition/health intervention can be found in Appendix D. Our "intensive" MI condition refers to our 9-session manual intervention. As detailed in the Preliminary Studies Section, the development of our manual, methods for stage 1 pilot testing, and procedures for training therapists have followed recommendations made by Rounsaville, Carroll, and Onken (2001) and Carroll et al. (2006). As a stage 2 behavioral trial, the study includes an assessment of dose-response relationships and has a high likelihood of illuminating potential mechanisms of action within a single data collection site. Positive findings here will lead to stage 3 applications examining the effectiveness of the intervention in community-based settings using multi-site designs that would allow broader generalization.

MA dependent participants will be recruited from the New Leaf outpatient treatment program in Lafayette, California. This data collection site has a history of successfully recruiting MA dependent clients into research protocols (e.g., Galloway, et. al., 2000; Rawson et. al., 2004). In addition to receiving one of the MI interventions, all participants will receive standard outpatient treatment offered at New Leaf.

The specific aims and hypotheses are detailed below. In addition to comparing treatment conditions on outcome measures, in an overlaid naturalistic design we will build upon MI research examining mediators of outcome conducted by Moyers, Miller & Hendickson (2005). We propose to assess the impact of a modified definition of feedback on the therapeutic alliance and in turn on MA use. Our definition of feedback includes providing objective information and personalized feedback to clients, but we add to this our construct of supportive confrontation (Polcin, 2006a; Polcin, Galloway & Greenfield, 2006; Polcin, Galloway, Bostrom & Greenfield, 2007; Polcin & Greenfield, 2006). This concept entails providing warnings to the client about potential harm that might result if action is not taken to address problem areas. Supportive confrontation is an integral part of feedback in our MI interventions and we provide data in our Preliminary Studies (see the Measuring Confrontation during Recovery subheading) indicating that this type of confrontation is experienced as supportive, accurate and helpful (e.g. Polcin et al., 2006). We also suggest that our findings are consistent with the work of Moyers, et al. (2005), who found some confrontational interventions were associated with an enhanced therapeutic alliance when they were delivered from therapists with a high degree of skill. To avoid destructive interactions that Miller, Benefield and Tonigan (1993) found to be counterproductive (e.g., argumentation) therapists will "roll with resistance" when encountering clients who react defensively or reject confrontational statements.

Aim 1. To compare MA use and retention in treatment among clients receiving intensive and standard MI.

Hypothesis 1.1: The intensive MI condition will demonstrate longer retention in treatment, fewer days of MA use, and fewer positive urine tests than the standard MI condition during the first 9 weeks of treatment.

Hypothesis 1.2: The intensive MI condition will demonstrate fewer days of MA use and fewer positive urine tests than the standard MI condition at the 2-, 4-, and 6-month follow-ups.

Aim 2. To compare Addiction Severity Index (ASI) scales among clients receiving intensive and standard MI.

Hypothesis 2.1: ASI scores for clients in the intensive condition will be significantly lower than scores in the standard condition at 2-, 4-, and 6-month follow-ups.

Aim 3. To assess whether feedback enhanced with supportive confrontation directly impacts outcome and impacts outcome indirectly through a stronger therapeutic alliance.

Hypothesis 3.1: Higher Frequency/Extensiveness and Skill Level of Feedback enhanced with supportive confrontation will decrease MA use.

Hypothesis 3.2: Higher Frequency/Extensiveness and Skill Level of Feedback enhanced with supportive confrontation will enhance the therapeutic alliance, which will in turn impact MA use.

Exploratory Analyses

1. We will make repeated measures comparisons between the two treatment conditions for use of alcohol and other drugs in addition to MA. These will include self-report measures as well as urine screens and breathalyzer results.
2. We will compare intensive and standard MI on services utilization, which assesses use of additional formal treatment and informal recovery services such as self-help groups.
3. We will compare longitudinal measures of motivation between the two conditions and assess whether higher motivation is associated with better outcome. 4) We will compare HIV risk behaviors among clients receiving intensive and standard MI.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old,
2. Meets DSM IV criteria for MA dependence during the past year as assesses by the DSM-IV Checklist,
3. able to speak and read English,
4. capable of giving informed consent, and
5. likely to be in the area the next 6 months.

Exclusion Criteria:

1. requires inpatient treatment for detoxification, medical or psychiatric treatment, and
2. Serious psychiatric condition that would impair their ability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2009-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Polcin, Ed.D., Principal Investigator — Alcohol Research Group / Public Health Institute
Locations (1):
- Alcohol Research Group, Emeryville, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD

REFERENCES:
- [Background] Burke BL, Arkowitz H, Menchola M. The efficacy of motivational interviewing: a meta-analysis of controlled clinical trials. J Consult Clin Psychol. 2003 Oct;71(5):843-61. doi: 10.1037/0022-006X.71.5.843. PMID 14516234
- [Background] Carroll KM, Ball SA, Nich C, Martino S, Frankforter TL, Farentinos C, Kunkel LE, Mikulich-Gilbertson SK, Morgenstern J, Obert JL, Polcin D, Snead N, Woody GE; National Institute on Drug Abuse Clinical Trials Network. Motivational interviewing to improve treatment engagement and outcome in individuals seeking treatment for substance abuse: a multisite effectiveness study. Drug Alcohol Depend. 2006 Feb 28;81(3):301-12. doi: 10.1016/j.drugalcdep.2005.08.002. Epub 2005 Sep 28. PMID 16169159
- [Background] Rawson RA, Marinelli-Casey P, Anglin MD, Dickow A, Frazier Y, Gallagher C, Galloway GP, Herrell J, Huber A, McCann MJ, Obert J, Pennell S, Reiber C, Vandersloot D, Zweben J; Methamphetamine Treatment Project Corporate Authors. A multi-site comparison of psychosocial approaches for the treatment of methamphetamine dependence. Addiction. 2004 Jun;99(6):708-17. doi: 10.1111/j.1360-0443.2004.00707.x. PMID 15139869
- [Background] Polcin DL, Galloway GP, Palmer J, Mains W. The case for high-dose motivational enhancement therapy. Subst Use Misuse. 2004 Jan;39(2):331-43. doi: 10.1081/ja-120028494. PMID 15061564
- [Background] Galloway GP, Polcin D, Kielstein A, Brown M, Mendelson J. A nine session manual of motivational enhancement therapy for methamphetamine dependence: adherence and efficacy. J Psychoactive Drugs. 2007 Nov;Suppl 4:393-400. doi: 10.1080/02791072.2007.10399900. PMID 18286727
- [Background] Martino S, Ball SA, Gallon SL, et al. Motivational Interviewing Assessment: Supervisory tools for enhancing proficiency Salem, OR: Northwest Frontier Addiction Technology Transfer Center, Oregon Health and Science University. 2006 [Accessed: 2013-02-05. Archived by WebCite® at http://www.webcitation.org/6EDD4BNKM];
- [Background] Moyers TB, Miller WR, Hendrickson SML. How does motivational interviewing work? Therapist interpersonal skill predicts client involvement within motivational interviewing sessions. J Consult Clin Psychol. 2005 Aug;73(4):590-598. doi: 10.1037/0022-006X.73.4.590. PMID 16173846
- [Background] Polcin DL. Reexamining confrontation and Motivational Interviewing. Addict Disord Their Treat 2006;5:201-9.
- [Background] Polcin DL, Brown M, Galloway GP. Intensive Motivational Enhancement Therapy Manual. Berkeley, CA: Alcohol Research Group; 2005.
- [Background] Rawson RA, Condon TP. Why do we need an Addiction supplement focused on methamphetamine? Addiction. 2007 Apr;102 Suppl 1:1-4. doi: 10.1111/j.1360-0443.2006.01781.x. PMID 17493048
- [Background] Anglin MD, Urada D, Brecht ML, Hawken A, Rawson R, Longshore D. Criminal justice itreatment admissions for methamphetamine use in California: a focus on Proposition 36. J Psychoactive Drugs. 2007 Nov;Suppl 4:367-81. doi: 10.1080/02791072.2007.10399898. PMID 18284103
- [Background] Vocci FJ, Appel NM. Approaches to the development of medications for the treatment of methamphetamine dependence. Addiction. 2007 Apr;102 Suppl 1:96-106. doi: 10.1111/j.1360-0443.2007.01772.x. PMID 17493058
- [Background] Harris MH. Meth--it's everybody's problem. S D J Med. 2003 Sep;56(9):375-6. No abstract available. PMID 14524136
- [Background] Galloway GP, Marinelli-Casey P, Stalcup J, Lord R, Christian D, Cohen J, Reiber C, Vandersloot D. Treatment-as-usual in the methamphetamine treatment project. J Psychoactive Drugs. 2000 Apr-Jun;32(2):165-75. doi: 10.1080/02791072.2000.10400225. PMID 10908004
- [Background] Miller WR, Benefield RG, Tonigan JS. Enhancing motivation for change in problem drinking: a controlled comparison of two therapist styles. J Consult Clin Psychol. 1993 Jun;61(3):455-61. doi: 10.1037//0022-006x.61.3.455. PMID 8326047
- See also: website — http://www.arg.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized using stratified permuted blocks to ensure balance by gender and meth severity (defined as 10 or more days of meth use in the past month vs. less than 10 days in the past month)
Pre-assignment Details: A total of 620 participants were screened for the study over the 36 month period with 563 meeting eligibility. Of the 563, 308 completed baseline assessments and 217 of them were randomized to an MI treatment condition; 91 persons completed a baseline interview but did not show up for randomization.
Groups:
- 9 Sessions of Motivational Interviewing: Respondents received 9 1-hour sessions of Motivational Interviewing therapy concurrent with outpatient drug treatment.
  Intensive Motivational Interviewing: Weekly individual therapy sessions over 9 weeks (Intensive MI condition) consisting of supportive and directive interventions. The control condition consists on a single session of MI and nutritional education.
- 1 Session of Motivational Interviewing + 8 Sessions Nutrition: Respondents received one 1.5-hour session of Motivational Interviewing therapy at the outset of entering outpatient drug treatment.
  Single session of Motivational Interviewing
Period: Overall Study
Arm/Group | 9 Sessions of Motivational Interviewing | 1 Session of Motivational Interviewing + 8 Sessions Nutrition
Started | 111 | 106
Completed | 104 | 97
Not Completed | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 9 Sessions of Motivational Interviewing | 1 Session of Motivational Interviewing + 8 Sessions Nutrition | Total
Number analyzed (Participants) | 111 | 106 | 217
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 111 | 105 | 216
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (9.7) | 38.9 (10.8) | 38.6 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 53 | 107
  Male | 57 | 53 | 110
Region of Enrollment [Number; unit: participants]
  United States | 111 | 106 | 217

OUTCOME MEASURES:

1. Primary Outcome: Methamphetamine Days of Abstinence : Proportion of Days Abstinent
Description: The proportion of days abstinent from methamphetamine was represented by univariate averages at each interview of the overall adjusted longitudinal treatment effects for each of the Standard (SMI) and Intensive (IMI) conditions. For example, a baseline average of 0.55 at baseline represents that study participants were abstinent, on average 55% of the days measured.
Time Frame: Weekly while in treatment (9 weeks) and 4 and 6 month follow up
Measure: Mean (Standard Error); unit: proportion of days abstinent
Arm/Group | 9 Sessions of Motivational Interviewing | 1 Session of Motivational Interviewing + 8 Sessions Nutrition
Number analyzed (Participants) | 111 | 106
proportion of days abstinent
  Baseline | .56 (.04) | .55 (.04)
  2 Months | .74 (.03) | .74 (.04)
  4 Months | .75 (.03) | .76 (.03)
  6 Months | .75 (.03) | .78 (.03)
Statistical Analysis 1: Comparison: 9 Sessions of Motivational Interviewing vs 1 Session of Motivational Interviewing + 8 Sessions Nutrition; Stat Mixed Model Estimated was: MI9 (Post - Bline) - MI1 (Post - Bline) taken across 2, 4, and 6 month follow-ups adjusted for gender, age, and # sessions attended. This was done because a statistical test of trend of the post-baseline effect across the 3 post interviews indicated a homogeneous post-baseline treatment effect across time for both MI1 and MI9 conditions; Test type: Superiority or Other; p = .47, Random Effects modeling; Time averaged post-bline diff in diff = -.006, 95% CI 2-sided [-.023 to .011] — Stat Mixed Model: MI9 (Post - Bline) - MI1 (Post - Bline) taken across 2, 4, and 6 month follow-ups adjusted for gender, age, and # sessions attended

2. Secondary Outcome: Addiction Severity Index
Description: Addiction Severity Index - Lite (ASI) is a standardized, structured interview that assesses past 30 days problem severity in seven areas. These seven areas include medical, employment, drug, alcohol, legal, family/social and psychiatric status. Problem severity is rated on a scale of 0.0 - 1.0 with a higher score indicative of more problem severity. All scales have a range from 0 to 1.0.
Time Frame: Baseline, 2-,4-, and 6-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | 9 Sessions of Motivational Interviewing | 1 Session of Motivational Interviewing + 8 Sessions Nutrition
Number analyzed (Participants) | 111 | 106
units on a scale
  Baseline | .27 (.01) | .26 (.01)
  2 Months | .22 (.01) | .19 (.01)
  4 Months | .19 (.01) | .17 (.01)
  6 Months | .18 (.01) | .18 (.01)
Statistical Analysis 1: Comparison: 9 Sessions of Motivational Interviewing vs 1 Session of Motivational Interviewing + 8 Sessions Nutrition; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .034, Random effects model; Time averaged post-bline diff in diff = .007, 95% CI 2-sided [.001 to .013] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Description: This was a psycho-social study and no pharmacological medications were introduced or administered. Participants were monitored for serious adverse events and other, non-serious events but none were observed.
Arm/Group | 9 Sessions of Motivational Interviewing | 1 Session of Motivational Interviewing + 8 Sessions Nutrition
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/106
Other Adverse Events (participants affected / at risk) | 0/111 | 0/106

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes